CLINICAL TRIAL: NCT06352021
Title: The Effect of Distraction With a Kaleidoscope on the Level of Perceived Pain During Blood Sampling in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: İlknur KAHRİMAN (Other)
Responsible Party: Sponsor-Investigator, İlknur KAHRİMAN, Associate Professor, Karadeniz Technical University
Organization: Karadeniz Technical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KAHRİMAN İlknur
Record Dates: First submitted 2024-03-17; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Pain
Keywords: Blood collection; Distraction; Non-pharmacological treatment; Pain; Schoolchild
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kaleidoscope group (Experimental): The children in the kaleidoscope group were shown the kaleidoscope by the researcher five minutes before the blood sampling, and they were encouraged to look at the kaleidoscope during the procedure and describe the patterns they saw.
  Interventions: Device: kaleidoscope
- control group (No Intervention): This group underwent routine blood sampling procedures and did not receive any intervention to reduce their pain.

INTERVENTIONS:
Device: kaleidoscope — The children in the kaleidoscope group were shown the kaleidoscope by the researcher five minutes before the blood sampling, and they were encouraged to look at the kaleidoscope during the procedure and describe the patterns they saw. All children in the Kaleidoscope group agreed to participate in the study. All children in the kaleidoscope group were asked to look at the kaleidoscope just before the tourniquet was placed on their arms before the blood sampling procedure and to describe the patterns, they saw in it by turning it slowly during the procedure.
  Arms: kaleidoscope group

SUMMARY:
This experimental study aimed to determine the effect of distracting children with a kaleidoscope during blood sampling on their perception of pain during the procedure and to increase and improve the quality of evidence for the effectiveness of these methods across different populations and cultures.

Hypothesis 0 (H0): There is no difference between the pain scores of the kaleidoscope group and the control group during blood sampling.

Hypothesis 1 (H1): There is a difference between the pain scores of the kaleidoscope group and the control group during blood sampling.

DETAILED DESCRIPTION:
A pain-free life is the right of every child. Eliminating pain and improving the quality of life of children is one of the main goals of nursing care. Pediatric nurses should choose the appropriate assessment tool for the child's age and developmental characteristics and diagnose pain correctly. For this purpose, nurses can use appropriate distraction methods. Since the nurse is the healthcare worker who is with the child and family the most throughout the day, s/he should closely monitor and evaluate the child's pain and inform the child and family about the principles of pain control. Many hospitals in Türkiye generally do not use any non-pharmacologic methods to reduce procedural pain. Given that distraction techniques are inexpensive and easy to use, and that reducing children's pain may reduce negative feelings towards future procedures, it is important to examine the effectiveness of such methods. In our study, a kaleidoscope, one of the methods of distraction to reduce pain during blood sampling in children, was used. A kaleidoscope is a game tool that helps distract the child's attention from procedural pain and shows the external image by reproducing it when viewed through it. This experimental study aimed to determine the effect of distracting children with a kaleidoscope during blood sampling on their perception of pain during the procedure and to increase and improve the quality of evidence for the effectiveness of these methods across different populations and cultures.

ELIGIBILITY:
Inclusion Criteria:

* were being 7-12 years of age
* not having an auditory or visual disability
* not taking analgesics in the last eight hours
* not having any pain caused by other reasons before the procedure
* having vascular access and blood sampling interventions

Exclusion Criteria:

* having physical or mental disability
* having any nerve damage

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
The Wong-Baker Pain Scale | 5 minutes
  The scale was developed by Wong and Baker (1981) to assess pain between the ages of 3-18 years. It has been reported in the literature that it accurately measures children's pain. The scale has numerical values according to each facial expression. The lowest and the highest values are 0 and 5. As the score on the scale increases, sensitivity to pain decreases, and as the score decreases, sensitivity increases.

CONTACTS AND LOCATIONS:
Overall Officials: Ilknur Kahriman, Assoc. Prof., Study Director — Karadeniz Technical University; Beyhan Turkan, Master, Principal Investigator — TRABZON KANUNI EDUCATION RESEARCH HOSPITAL
Locations (1):
- Karadeniz Technical University Health Application and Research Center Farabi Hospital, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No